CLINICAL TRIAL: NCT03534050
Title: Neuropsychological and Oncological Outcomes in Grade 2 or 3 Glioma Patients Undergoing Postoperative Modern Radiotherapy - A Prospective Follow-up Study
Brief Title: Neuropsychological and Oncological Outcomes in Grade 2 or 3 Glioma Patients Undergoing Postoperative Modern Radiotherapy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-9201B
Record Dates: First submitted 2018-04-02; First posted 2018-05-23 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-03

CONDITIONS: Glioma of Brain
Keywords: Glioma; Low-Grade Glioma (LGG); Neurobehavioral Assessments; Neurocognitive Functions (NCF); Radiation Therapy (RT); Hippocampus; Progression-Free Survival (PFS)
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postoperative adjuvant RT (Experimental): In this prospective observational study, all potentially eligible patients are clinically indicated for receiving postoperative adjuvant RT. Namely, partial cranial irradiation will be initiated within one month approximately after enrollment. Prescription dose will be 5000 - 6000 cGy in 25 - 30 fraction during 5 - 7 weeks.
  Interventions: Radiation: postoperative adjuvant RT

INTERVENTIONS:
Radiation: postoperative adjuvant RT

SUMMARY:
Background: Infiltrative low grade gliomas (LGGs) are the most common primary central nervous system malignancies excluding the highest grade glioma, glioblastoma multiforme. Craniotomy with maximal safe tumor resection is endeavored to achieve longer survivals in LGG patients. Unfortunately, due to the infiltrative nature of gliomas and the frequent tumor location in eloquent areas, gross total resection is usually not applicable. According to National Comprehensive Cancer Network 2015 guidelines, postoperative adjuvant radiation therapy (RT) is recommended for most adult patients with low-grade infiltrative LGGs in order to enhance local control and prolong progression-free survival (PFS), except those who are no older than 40 years of age and in whom maximal safe resection is not feasible. However, brain irradiation-related neurocognitive function (NCF) sequelae are potentially and indeed a concern which should not be ignored. In terms of the time course of cranial irradiation-induced NCF decline, it might vary considerably according to the specific domains which are selected to be measured. Early neurocognitive decline principally involve impairments of episodic memory, which has been significantly associated with functions of the hippocampus. This study thus aims to investigate the impact of partial brain irradiation with using contemporary radiotherapeutic techniques on neurocognitive performances, intracranial local control, and progression-free survival in patients with intracranial high-risk grade 2 or 3 gliomas.

Methods: Patients with intracranial high-risk low-grade or grade 3 gliomas will be enrolled to this study once postoperative adjuvant RT is recommended. All eligible and recruited patients should receive baseline functional brain MRI examination and baseline neurobehavioral assessment. Subsequently, partial cranial irradiation will be initiated within one month approximately after enrollment. Brain RT dose will be 5000 - 6000 cGy in 25 - 30 fraction during 5 - 7 weeks. Accordingly, a battery of neuropsychological measures, which includes 7 standardized neuropsychological tests (e.g., executive functions, verbal & non-verbal memory, working memory, and psychomotor speed), is used to evaluate neurobehavioral functions for our registered patients. The primary outcome measure is delayed recall, as determined by the change/decline in verbal memory or non-verbal memory from the baseline assessment to 4 months after the start of postoperative adjuvant RT.

ELIGIBILITY:
Inclusion Criteria:

* All patients with infiltrative low-grade gliomas who have received craniotomy plus tumor removal or at least biopsy with pathologic conformation; brain radiation therapy is recommended owning to some high-risk features including subtotal resection (STR) or age at craniotomy older than 40 years old
* Good performance status no worse than Eastern Cooperative Group (ECOG) of 2 or a general status of Karnofsky Score (KPS) at least 70 %

Exclusion Criteria:

* A pathological diagnosis confirmed to be WHO grade IV glioma (i.e., glioblastoma multiforme) or grade I disease (i.e., pilocystic astrocytoma)
* Radiographic evidence of gliomatosis cerebri
* Prior cranial irradiation for any reasons

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is delayed recall, as determined by the change/decline in verbal memory (WMS III- Word List score) from the baseline assessment to 4 months after the start of postoperative adjuvant RT. | 4 months after the start of postoperative adjuvant RT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in verbal memory [Wechsler Memory Scale - 3rd edition (WMS III) - Word List score] from the baseline assessment to 4 months after the start of the course of postoperative adjuvant RT.
The primary endpoint is delayed recall, as determined by the change/decline in non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of postoperative adjuvant RT. | 4 months after the start of postoperative adjuvant RT
  Neurocognitive assessment: including memory, executive functions, and psychomotor speed. This neurocognitive outcome was delayed recall, as determined by the change/decline in non-verbal memory (WMS III- Visual Reproduction score) from the baseline assessment to 4 months after the start of the course of postoperative adjuvant RT.

SECONDARY OUTCOMES:
Overall survival time, indicated by the time from the date of recruitment to the date of expiring. | up to 24 months
The time from the date of recruitment to that of intracranial progression/failure noted on brain MRI or CT. | up to 24 months
The delayed recall will follow up until 24 months after the start of postoperative adjuvant RT. | up to 24 months
  The follow-up of neurocognitive assessment will be administered at 8 months, 12 months, 18 months and up to 24 months after the start of postoperative adjuvant RT.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin SY, Chuang CC, Huang YC, Pai PC, Lee CC, Wei KC, Tseng CK, Yang CC. Neuropsychological performances in patients with infiltrative non-GBM gliomas after postoperative adjuvant photon or proton radiotherapy: A prospective and preliminary investigation. Appl Neuropsychol Adult. 2024 Jul-Aug;31(4):606-615. doi: 10.1080/23279095.2022.2048830. Epub 2022 Mar 27. PMID 35343323